CLINICAL TRIAL: NCT03330483
Title: Do Hydrophilic Catheters Decrease Pain and Discomfort of a Patient During Urodynamic Study: Single-blinded Randomized Study
Brief Title: Do Hydrophilic Catheters Decrease Pain and Discomfort of a Patient During Urodynamic Study
Acronym: HYDRUDS
Status: Terminated | Type: Observational
Why Stopped: Difficulty in recruiting patients
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0246-16-MMC
Record Dates: First submitted 2017-10-04; First posted 2017-11-06 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Pain; Discomfort
Keywords: pain; discomfort; hydrophylic catheter; urodynamic study
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Female Speedicath nelathon: Evaluation of pain or discomfort in female patients at/during/after Speedicath nelathon-tip catheter insertion
- Female nelathon: Evaluation of pain or discomfort in female patients at/during/after standard nelathon-tip catheter insertion
- Male Speedicath tiemann: Evaluation of pain or discomfort in male patients at/during/after Speedicath tiemann-tip catheter insertion
- Male tiemann: Evaluation of pain or discomfort in male patients at/during/after standard tiemann-tip catheter insertion

SUMMARY:
This study attempts to verify whether different types of catheters could impact on patients' feelings at the first-time catheter insertion at urodynamic study.

Each patient will undergo an insertion of only one type of a catheter and will rate his/her pain and discomfort feelings.

DETAILED DESCRIPTION:
Urodynamic study usually starts with non-invasive uroflowmetry following by insertion of a urethral catheter (nelathon or tiemann tip) for measuring of post-void residual of urine. Insertion of a urethral catheter is usually accompanied by a discomfort and sometimes even a pain. In order to minimize these unpleasant feelings urodynamic technician uses gel with anesthetic agents.

Single-use sterile catheters without any equipment and no coating can be used with lubricants and nowadays are the standard equipment at urodynamic study. Non-coated standard catheters are widely considered in the literature to cause an increase in urethral irritation, poor patient satisfaction, increased bacteriuria, and long-term urethral complications. Single-use sterile catheters with hydrophilic coatings, ready-to-use solution, with gel on the surface of the catheter or gel in the wrapping. Hydrophilic-coated catheters are characterized by having a layer of polymer coating, which absorbs and binds water to the catheter up to 10 times its own weight. This results in a thick, smooth and slippery surface reducing friction between the catheter surface and the urethral mucosa during insertion. The coating layer remains intact upon introduction into the urethra and ensures lubrication of the urethra in its entire length. Coloplast Speedicath hydrophylic catheters are designed for single use and are pre-coated to allow ease of insertion and removal, thereby reducing the risk of urethral mucosal irritation that can be more prevalent in an non-coated product.

Up today, there are no studies to verify whether a patient has different feelings with different type of catheters during the first-time urethral cauterization at urodynamic study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients
2. Age 18 and above
3. Scheduled and consented for urodynamic study
4. Able to sign an informed consent and agree to be included to a study.

Exclusion Criteria:

1. indwelling catheter
2. use of pain killers in 24 hours prior to urodynamic study
3. persistent abdominal, perineal or pelvic pain or discomfort prior to a study
4. prior or suspected urethral stricture
5. urinary tract infection
6. positive asymptomatic urine culture prior to urodynamic study
7. scheduled for a transurethral cystoscopic examination at the same day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred to Urodynamic Suite at Meir Medical Center and comply with inclusion criteria
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain and discomfort level from a baseline | 0, 2, 15, 30 minutes
  Change in Visual Analogue Scale (VAS) questionnaire score from a baseline. VAS questionnaire score assesses pain and discomfort of a patient from 0 to 10 where 0 is no pain and discomfort and 10 is a maximal pain and discomfort.

SECONDARY OUTCOMES:
Change in pulse rate | 0, 2, 15, 30 minutes
  Pulse rate/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No